CLINICAL TRIAL: NCT05137951
Title: Validity and Reliability of Rebee Wearable Sensor to Measure Knee Joint Range of Motion
Brief Title: Validity and Reliability of Rebee Sensor to Measure Knee ROM
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Ahmed Saleh, demonstrator of basic science faculty of physical therapy, Cairo University
Other Study IDs: Validity of rebee sensor (PT)
Record Dates: First submitted 2021-10-03; First posted 2021-11-30 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-11

CONDITIONS: Physical Therapy Modalities
Keywords: Rebee Sensor; Digital goniometer; Knee joint Range of motion

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Rebee sensor — Rebee is a wearable motion sensor package of sensor with its own mobile application, which measures range of joint movement in different planes easily which the patient able to wear the sensor and move easily to measure ROM and record the measurement at the application software Digital goniometer Goniometry has been described as a tool to measure angle. It gives the physician a useful method to diagnose musculoskeletal function in terms of ROM, monitor the progress of an intervention, record the data for future follow-up, and meet statutory and legal requirements for impairment rating and disability determinations where applicable
  Other Names: Digital goniometer

SUMMARY:
This study was conducted to investigate:

The criterion related validity of Rebee wearable sensor in measuring active flexion and extension of knee joint ROM compared with digital goniometer measurement.

The intra-rater reliability of Rebee wearable sensor in measuring active flexion and extension of knee joint ROM compared with digital goniometer measurement.

DETAILED DESCRIPTION:
Range of Motion (ROM) of the joint is one of the factors that determine function of the musculoskeletal system. This parameter should be measured and recorded by a valid and reliable method . It is considered to be an essential component of lower limb physical examination, which can be applied using various instruments such as goniometers and inclinometers .

Range of motion of the knee joint is one of the major factors determining the outcome after knee injuries. It is also an important measurement required by many knee scoring systems to determine the preoperative status and postoperative outcome .

Measurements are used by physical therapists to quantify limitations of motion, it used to decide an appropriate therapeutic interventions and document the effectiveness of these interventions. The ideal measuring device should give reproducible valid and reliable data .It is required an essential skill in the musculoskeletal assessments commonly performed by physiotherapists.

Two-arm digital goniometer is still widely used in measuring uniaxial ROM of the joint of extremity, there is high validity, intra- rater and inter-rater reliability of the digital goniometer. It is considered valid and reliable tool that simplify physical therapists' work .The digital goniometer is the most commonly utilized clinical tool for measuring joint range of motion, the evolution of sensors technology and applications are easy to use, relatively inexpensive, and highly accessible .

Rebee is a wearable motion sensor package of sensor with its own mobile application, which measures range of joint movement in different planes easily which the patient able to wear the sensor and move easily to measure ROM and record the measurement at the application software, that is facilitate the tele-measurement which the patients are supposed to put on the sensors and perform the actions themselves, or with assistance from physical therapist.

There is lack in the literature about using Rebee wearable sensor in measuring the range of knee joint so this study was conducted to test the criterion related validity and intrarater reliability of the rebee wearable sensor in measuring active knee joint ROM compared with digital goniometer measurement.

ELIGIBILITY:
Inclusion Criteria:

* Forty normal participant's age ranged from 30 to 45.
* The participant from both sex.
* Participant Body mass index (BMI) from (19 to 25) normal weight (BMI= weight (kg) / [height (m)] 2)

Ages: 30 Years to 45 Years | Sex: All
Age Groups: Adult
Study Population: The participants were recruited from Faculty, staff, and students of Pharos University, Alexandria, Egypt. Graduate Program in Physical Therapy after achieving the inclusion criteria .
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-25 (Actual)

PRIMARY OUTCOMES:
test Validation of rebee wearable sensor for measuring knee Range of motion | day 1
  The criterion related validity andof Rebee wearable sensor in measuring active flexion and extension of knee joint ROM compared with digital goniometer measurement.
test intrarater reliability of rebee wearable sensor to measure active knee flexion and extension ROM | day 1
  the procedures was repeated two times with one week interval between measurements. Researcher was recorded all the measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Wadida H Abd elkader, PhD, Study Director — Professor.dr
Locations (1):
- Pharos university at alexandria, Alexandria, Egypt

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-11-10): https://cdn.clinicaltrials.gov/large-docs/51/NCT05137951/Prot_SAP_ICF_000.pdf